CLINICAL TRIAL: NCT06239740
Title: Effects of Electroacupuncture on Cognitive Symptoms in Major Depressive Disorder: A Pilot Study and Randomized Controlled Trial
Brief Title: Effects of Electroacupuncture on Cognitive Symptoms in Major Depressive Disorder
Acronym: ELECACU-COG-Pi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Yindee Boontra, Doctor of Medicine, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTU-EC-PS-1-304/64; Thammasat University (Other: Faculty of Medicine, Thammasat University)
Record Dates: First submitted 2024-01-12; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorders; Cognitive Dysfunction
Keywords: Electroacupuncture; Depression; Cognition; Humans; Pilot; Randomized Controlled Trial
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction; Depression | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: In the electroacupuncture group (EG), participants received acupuncture at 10 scalp points (Baihui [GV20], Ex-hn 1, 3 points of intelligence [Shenting [GV24], Benshen [GB13] on both sides, Touwei [ST8] on both sides). Electroacupuncture was applied for 20 minutes at Benshen [GB13] and Touwei [ST8] on both sides. They also received acupuncture at Tai chong [LV3], Tai Yuan [LU9], and Tai Xi [KI3] on both sides, as shown in picture 1. Acupuncture sessions were weekly for 10 weeks.
  In the sham acupuncture control group (CG), participants received acupress or a brief needle insertion at He gu on both hands during the first and 10th weeks, marking the endpoint of the study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In the sham acupuncture control group (CG), participants received acupress or a brief needle insertion at He gu on both hands during the first and 10th weeks, marking the endpoint of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): In the electroacupuncture group (EG), participants received acupuncture at 10 scalp points (Baihui [GV20], Ex-hn 1, 3 points of intelligence [Shenting [GV24], Benshen [GB13] on both sides, Touwei [ST8] on both sides). Electroacupuncture was applied for 20 minutes at Benshen [GB13] and Touwei [ST8] on both sides. They also received acupuncture at Tai chong [LV3], Tai Yuan [LU9], and Tai Xi [KI3] on both sides, as shown in picture 1. Acupuncture sessions were weekly for 10 weeks.
  Interventions: Procedure: Electroacupuncture group
- Sham acupuncture (Sham Comparator): In the sham acupuncture control group (CG), participants received acupress or a brief needle insertion at He gu on both hands during the first and 10th weeks, marking the endpoint of the study
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Electroacupuncture group — The acupuncture needle was placed on the scalp at a Chinese traditional acupuncture point. Subsequently, a small electrode was attached to the needle. A minor amount of electricity runs through the electrode, producing a slight vibration or soft hum during the treatment.
  Other Names: electroacupuncture
  Arms: Electroacupuncture group
Procedure: Sham acupuncture — participants received acupress or a brief needle insertion at He gu on both hands during the first and 10th weeks, marking the endpoint of the study
  Arms: Sham acupuncture

SUMMARY:
The goal of this pilot Study and Randomized Controlled Trial is to investigate the impact of electroacupuncture on cognitive function, quality of life (QoL), and depression severity in patients with major depressive disorder (MDD).

The main question[s] it aims to answer are:

* Primary : electroacupuncture has the potential to treat subjective cognitive complaints and cognitive impairment in MDD outpatients
* Secondary : electroacupuncture has the potential to treat depressive in MDD outpatients The 60 participants will randomly be assigned to either the treatment group or the control group in a 1:1 ratio. The treatment group will undergo electroacupuncture (EA), while the control group will receive sham acupuncture within 10 weeks period.

Both groups will receive antidepressants with adjunctive medication (i.e., benzodiazepines, tricyclics, or antipsychotics) as the standard treatment. All participants will be assessed for executive functions and memory using specific cognitive tests, including the Trail Making Test B (TMT-B), Stroop Color and Word Test (SCWT), category delayed recall in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog), and subjective reports of concern regarding concentration, memory, problem-solving, learning, communication, and quality of life (QoL) concerns using the WHO Disability Assessment Schedule (WHODAS 2.0; sections D1.1-1.6 and H1-3), and depressive symptoms were assessed using the Thai-PHQ-9.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 55 years
* MDD diagnosed according to the DSM-5 or DSM-IV-TR criteria,
* low suicidal risk
* receiving treatment with antidepressants for at least 3 months from psychiatrists and psychiatric residents.
* Subjective cognitive symptoms from the screening using the Thai version of the Patient Health Questionnaire (Thai-PHQ-9).

Exclusion Criteria:

* severe cognitive deficits from traumatic brain injury, delirium, neurodevelopmental disorders, or intellectual disability;
* neurological disorders such as stroke, Parkinson's disease, epilepsy, or other brain lesions;
* severe medical conditions preventing lying down for 20 minutes;
* recent electroconvulsive therapy (ECT) within the last 6 months;
* Individuals with a pacemaker;
* visual or hearing impairment that could not be corrected with eyeglasses or hearing aids;
* severe MDD or scoring 20 points or more on the Thai-PHQ-9.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-24 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Trail making test B (TMT-B) | Pre-intervention at the beginning point (T0) and the endpoint will be the 10th week (T10)
  The TMT- B is scored based on the time (in seconds) it takes to complete the test, including corrections for errors prompted by the examiner. A shorter time implies better performance.
The Stroop Color and Word Test (SCWT) | Pre-intervention at the beginning point (T0) and the endpoint will be the 10th week (T10)
  SCWT used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute."Score" refers to the number of words achieved, and a higher number of words indicates a better score.
ADAS-cog category delayed recall | Pre-intervention at the beginning point (T0) and the endpoint will be the 10th week (T10)
  ADAS-cog category delayed recall is used to assess memory. The score reflects the number of words that can be remembered. The more words remembered, the better the score.
Subjective cognitive complaint | Pre-intervention at the beginning point (T0) and the endpoint will be the 10th week (T10)
  WHODAS 2.0; sections D1.1-1.6 and H1-3, which is a questionnaire asking about the number of days in the past 30 days when participants experienced difficulties with attention, understanding, and initiating conversation. "Score" is the rating of the number of days with issues, and a decrease in score indicates improvement or a better outcome.

SECONDARY OUTCOMES:
Thai Patient Health Questionnaire (PHQ-9) | Pre-intervention at the beginning point (T0) and the endpoint will be the 10th week (T10)
  The Thai PHQ-9 (Patient Health Questionnaire-9) objectifies and assesses degree of depression severity via questionnaire. A lower score means better."

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The data set will be share on Zenodo
Supporting Information: Study Protocol
Time Frame: January 15, 2024 and for 5 years (Jan 14, 2029)
Access Criteria: no limitation
URL: https://doi.org/10.5281/zenodo.10488186

REFERENCES:
- [Derived] Boontra Y, Thanetnit C, Phanasathit M. Effects of electroacupuncture on cognitive symptoms in major depressive disorder: a pilot study and randomized controlled trial. F1000Res. 2024 Dec 23;13:479. doi: 10.12688/f1000research.146897.4. eCollection 2024. PMID 39620153
- Available data/document: Study Protocol — https://doi.org/10.5281/zenodo.10488186